CLINICAL TRIAL: NCT00005956
Title: A Pilot Study of Active Immunotherapy With HER2/Neu Intracellular Domain (ICD) Protein-Pulsed, Autologous, Cultured Dendritic Cells in Patients With No Evidence of Disease After Standard Treatment for HER2/Neu Expressing Malignancies
Brief Title: Biological Therapy in Treating Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1309; 6542 (Other: FDA); 1528 (Other: DUMC IRB); CDR0000067937 (Other: NCI)
Record Dates: First submitted 2000-07-05; First posted 2003-05-21 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer; Gastric Cancer; Ovarian Cancer
Keywords: stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; stage IIIB breast cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: HER-2/neu intracellular domain protein
  Other Names: HER2 ICD
Biological: therapeutic autologous dendritic cells
  Other Names: DC

SUMMARY:
RATIONALE: A person's white blood cells mixed with tumor proteins may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of biological therapy in treating patients who have advanced cancer that shows no signs of disease following treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the immune response of patients with HER2/neu expressing advanced malignancies showing no evidence of disease after standard treatment when injected with HER2/neu intracellular domain protein pulsed autologous dendritic cells.
* Assess time to recurrence in these patients.

OUTLINE: Autologous dendritic cells (DC) are pulsed with HER2/neu intracellular domain protein (ICD). The pulsed DC are administered subcutaneously (SQ) and intradermally, followed by autologous DC mixed with tetanus toxoid (TT) and autologous DC mixed with keyhole limpet hemocyanin (KLH) SQ and intradermally on day 1. HLA-A2 positive patients also receive autologous DC mixed with CMV pp65 peptide SQ and intradermally on day 1. Treatment continues every 3 weeks for a total of 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year or until disease progression.

PROJECTED ACCRUAL: A total of 6 patients will be accrued for this study over 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced malignancy that expresses HER2/neu

  * Stage IIA breast cancer with more than 6 positive lymph nodes
  * Stage IIB, IIIA, or IIIB breast cancer
  * Stage III ovarian cancer
  * Lymph node positive gastric cancer
  * Metastatic tumor
* No measurable or evaluable disease after standard treatment
* No previously irradiated or newly diagnosed CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Menopausal status:

* Not specified

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Greater than 6 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Hemoglobin at least 9 mg/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* No hepatic disease, including viral hepatitis

Renal:

* Creatinine less than 2.5 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Pulmonary:

* No asthma or chronic obstructive pulmonary disease

Immunologic:

* Must have positive intradermal delayed hypersensitivity test for at least 1 of the following:

  * Candida
  * Mumps
  * Tetanus
  * Trichophyton
  * Histoplasmin
* No prior autoimmune disease including, but not limited to, the following:

  * Inflammatory bowel disease
  * Systemic lupus erythematosus
  * Ankylosing spondylitis
  * Scleroderma
  * Multiple sclerosis

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* Hepatitis B surface antigen and hepatitis C antibody negative
* No other concurrent serious chronic or acute illness or infection (including urinary tract infection)
* No known shellfish or iodine allergy
* No other prior or concurrent malignancy except for nonmelanoma skin cancer, cervical cancer, or controlled superficial bladder cancer
* No medical or psychological condition that may preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No other concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy

Endocrine therapy:

* Concurrent hormonal therapy allowed (tamoxifen, raloxifene, toremifene, and all aromatase inhibitors)
* At least 4 weeks since prior steroid or immunosuppressive therapy (e.g, azathioprine or cyclosporine)

Radiotherapy:

* Prior radiotherapy allowed except to cranium
* At least 4 weeks since prior radiotherapy and recovered
* At least 12 weeks since prior strontium chloride Sr 89
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior surgery and recovered

Other:

* Concurrent bisphosphonates allowed
* No prior hepatitis B immunization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2000-02; Primary Completion 2001-08 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months
  safety

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Morse, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Morse MA, Hobeika A, Osada T, Niedzwiecki D, Marcom PK, Blackwell KL, Anders C, Devi GR, Lyerly HK, Clay TM. Long term disease-free survival and T cell and antibody responses in women with high-risk Her2+ breast cancer following vaccination against Her2. J Transl Med. 2007 Sep 6;5:42. doi: 10.1186/1479-5876-5-42. PMID 17822557